CLINICAL TRIAL: NCT05261542
Title: Detection of Cancer Cells and Tumor Margins During Colorectal Cancer Surgery by Intraoperative Flow Cytometry
Brief Title: Intraoperative Flow Cytometry In Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: University Hospital, Ioannina (Other)
Responsible Party: Principal Investigator, CHRISTINA BALI, ACCOSIATE PROFESOR OF SURGERY, University Hospital, Ioannina
Other Study IDs: 27190/26-10-2017
Record Dates: First submitted 2022-02-06; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue samples from normal and cancer epithelium collected following colectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal colorectal epithelium: Tissue samples from normal colorectal epithelium are collected during colectomy in every colorectal cancer patient
  Interventions: Diagnostic Test: flow cytometry
- cancer colorectal epithelium: Tissue samples from colorectal cancer are collected during colectomy in every colorectal cancer patient
  Interventions: Diagnostic Test: flow cytometry

INTERVENTIONS:
Diagnostic Test: flow cytometry — evaluation of intraoperative flow cytometry in detecting cancer cells in colorectal epithelium

SUMMARY:
This study was designed to investigate the efficacy of flow cytometry to accurately identify between normal and cancer cells in colon epithelium in humans diagnosed with colorectal cancer.

DETAILED DESCRIPTION:
Tissue samples from normal and cancerous colon epithelium are collected intraoperatively following standard colectomy and analyzed blindly by flow cytometry, which reports, in less than 10 min, on the origin of the sample based in the estimation of DNA and tumor index.

ELIGIBILITY:
Inclusion Criteria:

biopsy proven colorectal cancer signed informed consent for participation

Exclusion Criteria:

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with colorectal cancer and being treated by standard colectomy or/and neoadjuvant theraphy according to current guidelines.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Accuracy of intraoperative Flow Cytometry for cancer cell identification in colorectal cancer. | 2017-2021
  Samples from cancer and normal colon epithelium are prospectively collected intraoperatively and assessed with intraoperative Flow Cytometry. Following comparative DNA content and phenotypic analysis, the receiver operating characteristic (ROC) curve analysis is used to evaluate the performance of intraoperative Flow Cytometry to distinguish between normal and cancer tissue. The optimal cut-off value is determined to delineate the status of tumor tissue, resulting in the highest sensitivity and specificity and hence the optimal accuracy.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ioannina, Ioannina, Epirus, Greece

IPD SHARING:
Plan to Share IPD: Undecided